CLINICAL TRIAL: NCT05345912
Title: A Randomized, Double Blind, Placebo-controlled, Dose-escalation, Crossover Study to Compare and Evaluate the Pharmacokinetics and Safety of 'CG-745 IV' Intravenous Formulation and 'CG-750' Capsule Formulation in Healthy Male Adults
Brief Title: Pharmacokinetics and Safety of 'CG-745 IV' and 'CG-750' in Healthy Male Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CrystalGenomics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CG200750-1-01
Record Dates: First submitted 2019-12-03; First posted 2022-04-26 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Healthy
MeSH Terms: interventions — N1-(3-(dimethylamino)propyl)-N8-hydroxy-2-((naphthalene-1-loxy)methyl)oct-2-enediamide; Saline Solution

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind, placebo-controlled, dose-escalation, crossover study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Subjects received 125 mg of either placebo IV or CG-745 IV infusion over 60 min. After 14 days wash-out period, subjects received 125 mg of either placebo (PO) or CG-750 capsule orally in the fasted state for at least 10 hours.
  Interventions: Drug: CG-745 IV Solution; Drug: CG-750 125mg capsule; Other: PO Placebo; Other: IV Placebo: 0.9 % normal saline
- Cohort 2 (Experimental): Subjects received 250 mg of either placebo IV or CG-745 IV infusion over 60 min. After 14 days wash-out period, subjects received 375 mg of either placebo (PO) or CG-750 capsule orally in the fasted state for at least 10 hours.
  Interventions: Drug: CG-745 IV Solution; Drug: CG-750 125mg capsule; Other: PO Placebo; Other: IV Placebo: 0.9 % normal saline
- Cohort 3 (Experimental): Subjects received 125 mg of either placebo IV or CG-745 IV infusion over 60 min. After 14 days wash-out period, subjects received 750 mg of either placebo (PO) or CG-750 capsule orally in the fasted state for at least 10 hours.
  Interventions: Drug: CG-745 IV Solution; Drug: CG-750 125mg capsule; Other: PO Placebo; Other: IV Placebo: 0.9 % normal saline

INTERVENTIONS:
Drug: CG-745 IV Solution — CG-745 IV: Supplied as 125 mg/vial Administered intravenously, once, approximately 9 AM local time in fasted condition, over 60 min infusion
  Other Names: CG200745
Drug: CG-750 125mg capsule — CG-750 capsule: Supplied as 125 mg/capsule Administered orally, once, approximately 9 AM local time in fasted condition except for fed condition in Cohort 2, period 3
  Other Names: CG200750
Other: PO Placebo — PO Placebo: Supplied as placebo capsule (same appearance as in CG-750 Administered orally, once, approximately 9 AM local time in fasted condition except for fed condition in Cohort 2, period 3
Other: IV Placebo: 0.9 % normal saline — IV Placebo: 0.9 % normal saline Administered intravenously, once, approximately 9 AM local time in fasted condition, over 60 min infusion

SUMMARY:
A randomized, placebo-controlled, dose-escalation, crossover study.

DETAILED DESCRIPTION:
Total of 24 health volunteers will be randomized to receive either of Cohort 1,2 or 3. (8 subjects each)

[Cohort 1] Subject will fast for at least 10 hours in first treatment, and then be administrated with CG-745 IV or placebo. After 2-week rest period, subject will fast for at least 10 hours in second treatment, and then be administrated CG-750 capsule or placebo with 150 mL of water.

[Cohort 2] The recommended dose of capsule in cohort 2 will be determined based on the bioavailabilty and safety data of cohort 1.

Subject will fast for at least 10 hours in first treatment, and then be administrated with CG-745 IV or placebo. After 2-week rest period, subject will fast for at least 10 hours in second treatment, and then be administrated the determined dose of CG-750 capsules or placebo with 150 mL of water.

After 2-week rest period, subject will take the high fat diet and then be administrated the determined dose of CG-750 or placebo with 150 mL of water.

[Cohort 3] The recommended dose of capsule in cohort 3 will be determined based on the bioavailabilty of cohort 1 and 2.

Subject will fast for at least 10 hours in first treatment, and then be administrated with CG-745 IV or placebo. After 2-week rest period, subject will fast for at least 10 hours in second treatment, and then be administrated the determined dose of CG-750 or placebo with 150 mL of water.

ELIGIBILITY:
Key Inclusion Criteria:

* Subject who signed voluntarily the written agreement after understanding the purpose, contents, the properties and expected adverse effects of investigational product
* Subject who is considered to be appropriate for the study according to the judgment of investigator based on physical examination, clinical laboratory test, electrocardiogram, vital sign and questionnaire

Key Exclusion Criteria:

* Subject with clinically meaningful and relevant disease in liver, kidney, nervous system, respiratory system, endocrine system, blood and tumor, cardiovascular system, urinary system and mental system
* Subject with sensitive reaction in HDAC inhibitor or another drug
* Subject who participated in another clinical trial or bioequivalent study with past 6 weeks
* Subject who is not considered to be appropriate for the study according to the judgment of investigator

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-12-16 (Actual); Primary Completion 2020-09-18 (Actual); Study Completion 2021-05-19 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration of CG200745 (Cmax) | 0 (pre-dose), 0.33 (20 min), 0.67 (40 min), 1 (60 min), 1.083 (1h 5 min), 1.25 (1h 15 min), 1.5, 2,3,4,5,6,7,9,12,25,48,72hr after dose
  Plasma level vs. time profiles were plotted for each subject in linear or log/linear graphs.
Area Under the Concentration-Time Curve (AUC 0-72h) | 0 (pre-dose), 0.33 (20 min), 0.67 (40 min), 1 (60 min), 1.083 (1h 5 min), 1.25 (1h 15 min), 1.5, 2,3,4,5,6,7,9,12,25,48,72hr after dose
  Plasma level vs. time profiles were plotted for each subject in linear or log/linear

SECONDARY OUTCOMES:
The Number of Participants Who Experienced Serious or Non-Serious Adverse Events | Up to 4 weeks for each dosing cohort

CONTACTS AND LOCATIONS:
Overall Officials: SeungHwan Lee, Ph.D, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea